CLINICAL TRIAL: NCT01907126
Title: HIV/STI Risk Reduction for Incarcerated Women With Interpersonal Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Jennifer Johnson, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH094188 (NIH); R34MH094188 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-07-24 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Unsafe Sex; Physical Violence; Sexual Assault; Sexual Abuse
Keywords: HIV; Sexually transmitted infections; Sexual abuse; Physical abuse; Women; Prison
MeSH Terms: conditions — Unsafe Sex; Sexually Transmitted Diseases | interventions — Food Assistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women's Prison CoOp (WPC) (Experimental): Will receive 5 group psychoeducation sessions plus individual pre-release and post-release goal planning sessions. Psychoeducation sessions will cover HIV risk and violence prevention, interpersonal violence-specific sexual safety skills, empowerment through knowledge and treatment, and skills for increasing affect regulation and social support.
  Interventions: Behavioral: Women's Prison CoOp (WPC)
- Nutrition program (NP) (Placebo Comparator): Participants in this condition will receive dose-matched nutrition education.
  Interventions: Behavioral: Nutrition Program (NP)

INTERVENTIONS:
Behavioral: Nutrition Program (NP) — Nutrition Program (NP) participants will receive the same number, format, and schedule of group and individual 60-minute sessions, which will focus on low-cost strategies for improving nutrition.
  Arms: Nutrition program (NP)
Behavioral: Women's Prison CoOp (WPC) — Weekly as 60-minute sessions, 3 group and two individual sessions during incarceration as close to prison discharge as possible. Session 1 focuses on understanding and reviewing HIV risks, including interpersonal violence. Session 2 addresses gender, power, violence, and affect management to counter the emotional effects of violence. Session 3 addresses IV-specific sexual safety skills, including affect management skills. Session 4 helps women begin to develop a personalized safety plan, which may include increasing social support and access to resources. Session 5 helps her finalize and practice the plan, and Session 6 problem-solves any difficulties that have arisen in executing the plan.
  Arms: Women's Prison CoOp (WPC)

SUMMARY:
The pilot study aims to conduct a randomized pilot trial in a sample of 40 incarcerated women with lifetime interpersonal violence who are 6-10 weeks away from release to demonstrate the feasibility and acceptability of the proposed recruitment methods and research design, of the intervention training methods, of delivering the enhanced Women's Coop and nutrition control interventions. Per recent guidance from NIMH, the investigators will also examine 95% confidence intervals around differences between the proposed intervention and a dose-matched control condition (Nutrition Program), for the following outcomes through 8 months post prison release: reduced unprotected vaginal or anal sex occasions and fewer cases of vaginal trichomoniasis (primary); reduced interpersonal violence episodes, symptoms of PTSD and depression, and drug using/heavy drinking days (secondary); and increased affect management and social support (including effectiveness in obtaining substance use, mental health treatment and other resources) (tertiary).

ELIGIBILITY:
Inclusion Criteria:

* Females in prison
* Experienced lifetime interpersonal violence (includes physical or sexual assault or abuse)
* At least one unprotected sexual occasion with a male partner within the 90 days prior to incarceration
* Approximately 6-10 weeks before release
* Expect to be released to locations within RI or MA

Exclusion criteria:

* Cannot complete intake interview due to problems with reality testing, brain impairment, or language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Unprotected Sexual Occasions (USOs; Vaginal and Anal) | Slope over time: Baseline, 2 months after release, 5 months after release, 8 months after release
  The investigators will calculate effect sizes and confidence intervals for number of USOs. The number of USOs will be measured by the Timeline Follow Back (TLFB).
Presence of Trichomoniasis | Slope over time: Baseline, 2 months after release, 5 months after release, 8 months after release
  The investigators will calculate odds ratios and 95% confidence intervals for any positive trichomoniasis test during follow-up using logistic regression, with baseline trichomoniasis status as a covariate. The presence of Trichomoniasis is measured by rapid test.
Treatment Acceptability | 2 months post release
  The investigators will assess the feasibility and acceptability of WPC and NP by examining rates of treatment attendance, rates of treatment completion (attending at least 5 of the 6 scheduled individual sessions) and drop-out, and scores on the End of Treatment Questionnaire. Additionally, they will examine reasons for termination for consistent patterns. Acceptability of both WPC and NP using data from Client Satisfaction Questionnaire and detailed exit interviews will be examined.
Treatment Feasibility | 2 months post release
  One of the primary goals of a treatment development study is to demonstrate the feasibility of the proposed treatment and of the study and recruitment methods. As a result, the investigators will assess the feasibility of the research procedures by examining study recruitment and refusal rates, participants' willingness to be randomized, follow-up rates, reliability and range of responses to study questionnaires, and success of the interventionist training program

SECONDARY OUTCOMES:
Interpersonal violence (IPV) episodes | Slope over time: Baseline, 2 months after release, 5 months after release, 8 months after release
  Episodes of interpersonal violence (physical or sexual abuse or assault) as measured by the Trauma History Questionnaire (THQ) and the Conflict Tactic Scale (CTS2). The investigators will calculate the effect size and 95% confidence intervals for number of interpersonal violence episodes during the follow-up period using Trauma History Q data. For women who have been in at least one romantic relationship during the follow-up period, the investigators will also explore differences in IPV severity using CTS2 scores. Exploratory tests for differences between conditions will use hierarchical linear modeling (HLM), with baseline scores as covariates.
PTSD Symptom Severity | Slope over time: Baseline, Pre-release, 2 months after release, 5 months after release, 8 months after release
  PTSD Symptom Severity as measured by the Davidson Trauma Scale (DTS). The investigators will calculate effect sizes and 95% confidence intervals for reduction in PTSD symptoms using the DTS total scores. Exploratory tests for differences between conditions will use HLM with baseline scores as covariates.
Depressive Symptom Severity | Slope over time: Baseline, Pre-release, 2 months after release, 5 months after release, 8 months after release
  Depressive Symptom Severity as measured by the Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR). The investigators will calculate effect sizes and 95% confidence intervals for reduction in depressive symptoms using the QIDS-SR total scores. Exploratory tests for differences between conditions will use HLM with baseline scores as covariates.
Post Release Drug Using/Heavy Drinking Days | Slope over time: 2 months after release, 5 months after release, 8 months after release
  Total number of days that women used drugs or had 4+ drinks as measured by the Timeline Followback (TLFB). Self-report data will be compared to significant other report, urine drug screens, and breath alcohol tests. The investigators will calculate effect sizes and 95% confidence intervals for number of drug using/heavy drinking days using TLFB data. Exploratory tests for differences bet-ween conditions will use HLM with using/heavy drinking days in the 90 prior to incarceration as a covariate

OTHER OUTCOMES:
Affect Management | Slope over time: Baseline, Pre-release, 2 months after release, 5 months after release, 8 months after release
  Affect management is measured by the Distress Tolerance Scale (DTS). It is a 15-item self report measure that assesses perceived ability to tolerate emotional distress, including ability to regulate negative affect. The investigators will calculate effect sizes and 95% confidence intervals for improvement in affect modulation measured by the DTS. Exploratory tests for differences between conditions will use HLM with the baseline score as a covariate.
Perceived Social Support | Slope over time: Baseline, Pre-release, 2 months after release, 5 months after release, 8 months after release
  Multidimensional Scale of Perceived Social Support (MSPSS) will be used to measure general social support. The investigators will calculate effect sizes and 95% confidence intervals for improvement in social support measured by the MSPSS using HLM with baseline score as a covariate.
Effectiveness in Obtaining Resources (EOR) and Treatment Received | Slope over time: Baseline, Pre-release, 2 months after release, 5 months after release, 8 months after release
  The Effectiveness in Obtaining Resources Scale assesses respondents' effectiveness in obtaining resources in 13 areas: housing, material, goods and services, education, employment, health care for themselves and their children, child care, transportation, social support, legal assistance, financial issues, and other issues regarding themselves and their children. For this study, the investigators also ask questions assessing a woman's ability to access mental health treatment, substance use, and partner violence resources. The Treatment Services Review (TSR) assesses receipt of mental health and substance use services.
  The investigators will also calculate effect sizes and 95% confidence intervals for effectiveness in obtaining resources measured by the EOR total score and for total days of treatment received measured by the TSR. Exploratory tests for differences between conditions will use HLM.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Johnson, PhD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Massachusetts CorrectionalInstitution - Framingham, Framingham, Massachusetts
  - South Middlesex CorrectionalCenter, Framingham, Massachusetts
  - Adult Correctional Institution, Cranston, Rhode Island

REFERENCES:
- [Derived] Kuo CC, Rosen RK, Zlotnick C, Wechsberg WM, Peabody M, Johnson JE. Sexual health prevention for incarcerated women: eroticising safe sex during re-entry to the community. BMJ Sex Reprod Health. 2018 Jun 28:bmjsrh-2017-200024. doi: 10.1136/bmjsrh-2017-200024. Online ahead of print. PMID 29954877